CLINICAL TRIAL: NCT04094896
Title: TCHP (Docetaxel/Carboplatin/Trastuzumab/Pertuzumab) Versus EC -THP(Epirubicin/ Cyclophosphamide Followed by Docetaxe/Trastuzumab/Pertuzumab) as Neoadjuvant Treatment for HER2-Positive Breast Cancer
Brief Title: TCHP Versus EC -THP as Neoadjuvant Treatment for HER2-Positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, KunWang, Professor, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018396H
Record Dates: First submitted 2019-09-17; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: HER2-Positive Breast Cancer
Keywords: Neoadjuvant Treatment; HER2-Positive Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: TCHP (Experimental): docetaxel/carboplatin/trastuzumab/Pertuzumab
  Interventions: Drug: TCHP
- Arm B: EC-THP (Active Comparator): epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab/Pertuzumab
  Interventions: Drug: TCHP

INTERVENTIONS:
Drug: TCHP — Both TCHP (docetaxel/carboplatin/trastuzumab/Pertuzumab) and EC followed by THP(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab/Pertuzumab)regimens as Neoadjuvant Treatment for HER2-Positive Breast Cancer have been recommended by NCCN guideline. It is unknown which regimen is better. This study is to evaluate the efficacy and safety ofTCHP (docetaxel/carboplatin/trastuzumab/Pertuzumab) and EC followed by THP(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab/Pertuzumab)regimens as Neoadjuvant Treatment in HER2- Positive breast cancer. The endpoint of pathologic complete response is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.
  Other Names: TCHP vs EC-THP

SUMMARY:
This study is to evaluate the efficacy and safety ofTCHP (docetaxel/carboplatin/trastuzumab/Pertuzumab) and EC followed by THP(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab/Pertuzumab)regimens as Neoadjuvant Treatment in HER2- Positive breast cancer. The endpoint of pathologic complete response is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.

DETAILED DESCRIPTION:
Both TCHP (docetaxel/carboplatin/trastuzumab/Pertuzumab) and EC followed by THP(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab/Pertuzumab)regimens as Neoadjuvant Treatment for HER2-Positive Breast Cancer have been recommended by NCCN guideline. It is unknown which regimen is better. This study is to evaluate the efficacy and safety ofTCHP (docetaxel/carboplatin/trastuzumab/Pertuzumab) and EC followed by THP(epirubicin/cyclophosphamide followed by docetaxe plus trastuzumab/Pertuzumab)regimens as Neoadjuvant Treatment in HER2- Positive breast cancer. The endpoint of pathologic complete response is used as a surrogate marker for survival. Safety and tolerability assessed by number of grade 4 toxicities and hospitalizations.

ELIGIBILITY:
Inclusion Criteria:

* • Histologically or cytologically confirmed HER2 positive invasive breast carcinoma

  * Clinical stage #-#B
  * Patients must have measurable disease as defined by palpable lesion with both diameters ≥2cm measurable with caliper and/or a positive mammogram or ultrasound with at least one dimension ≥2cm. Bilateral mammogram and clip placement is required for study entry. Baseline measurements of the indicator lesions must be recorded on the Patient Registration Form. To be valid for baseline, the measurements must have been made within the 14 days if palpable. If not palpable, a mammogram or MRI must be done within 14 days. If palpable, a mammogram or MRI must be done within 2 months prior to study entry. If clinically indicated, xrays and scans must be done within 28 days of study entry.
  * Eastern Cooperative Oncology Group(ECOG) performance status 0 to 1 within 14 days of study entry
  * Normal (greater than 50%) left ventricular ejection fraction (LVEF) by echocardiography
  * Signed informed consent
  * Adequate organ function within 2 weeks of study entry:

Absolute neutrophil count >1500/mm3, Hgb >9.0 g/dl and platelet count >100,000/mm3 Total bilirubin < upper limit of normal Creatinine < 1.5 mg/dL or calculated cranial cruciate ligament (CrCL) >50mL/min using the Cockcroft Gault equation serum glutamate oxaloacetate transaminase(SGOT)(AST) or serum glutamic oxaloacetic transaminase(SGPT)(ALT) and Alkaline Phosphatase must be within the range allowing for eligibility

* Patients must be over 18 years old.
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation.

Exclusion Criteria:

* • Metastatic disease

  * Prior chemotherapy, hormonal therapy, biologic therapy, investigational agent, targeted therapy or radiation therapy for current breast cancer. Patients with history of breast cancer greater than 5 years from initial diagnosis are eligible for the study. Patients may not have received anthracycline-based chemotherapy in the past. Patients with history of ductal carcinoma in situ(DCIS) are eligible if there were treated with surgery alone.
  * History of previous or current malignancy at other sites with the exception of adequately treated carcinoma in-situ of the cervix or basal or squamous cell carcinoma of the skin. Patients with a history of other malignancies, who remain disease free for greater than five years are eligible.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-09-17 (Actual); Primary Completion 2022-09-17 (Estimated); Study Completion 2022-09-17 (Estimated)

PRIMARY OUTCOMES:
pCR | one year
  pathologic complete response

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong General Hospital, Guangzhou, China